CLINICAL TRIAL: NCT06024447
Title: Impact of Subgingival Instrumentation on Masticatory Performance and Psychological Distress in Periodontitis: Stage III and IV
Brief Title: Impact of Subgingival Instrumentation on Masticatory Performance and Psychological Distress
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JANVIPERIO2023
Record Dates: First submitted 2023-08-10; First posted 2023-09-06 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stage III and Stage IV Periodontitis (Other): Subgingival Instrumentation will be performed in patients with Stage III and Stage IV periodontitis.
  Interventions: Procedure: Subgingival Instrumentation

INTERVENTIONS:
Procedure: Subgingival Instrumentation — Subgingival Instrumentation will be performed in patients with Stage III and IV periodontitis.

SUMMARY:
Patients of Stage III and Stage IV Periodontitis will be assessed for masticatory dysfunction and psychological distress. Subgingival Instrumentation will be done for treating periodontitis. Patients will be re-evaluated after 2 and 3 months in order to assess any change in masticatory dysfunction and psychological distress by improved periodontal health.

DETAILED DESCRIPTION:
Literature reveals that there occurs masticatory dysfunction in patients with Stage III and IV Periodontitis. It has been hypothesized that masticatory dysfunction along with halitosis and aesthetics of the patient can have an effect on the psychological distress in a chronic state.

Patients of Stage III and Stage IV Periodontitis with the following criteria will be included :

1. Adult patients with age group 30-50 years diagnosed with stage III/IV generalized periodontitis.
2. Presence of minimum 20 teeth (Eichner group A1, A2, A3) excluding third molars.

Exclusion Criteria: Patients with

1. Systemic diseases that may affect periodontal disease progression or outcome of treatment (diabetes, autoimmune diseases)
2. Systemic diseases that may affect masticatory ability of the patient (sarcopenia, TMJ disorders, Xerostomia, Acute Pulpitis)
3. History of periodontal treatment within the 6 months
4. Patients wearing orthodontic appliances
5. Diagnosed psychiatric disorder
6. History of antibiotic use within the previous 3 months
7. History of use of Steroid, immunosuppressive and psychiatric drugs
8. Pregnant and lactating women
9. Smoking or substance abuse
10. History of Menopause

Periodontal clinical parameters:

Plaque Index, Gingival Index, Bleeding on Probing, Probing Pocket Depth, Clinical Attachment Level, Mobility Psychological Parameters: Hospital Anxiety and Depression Scale -14 and Depression Anxiety and Stress Scale -21 Quality of Masticatory Dysfunction Questionnaire and Objective evaluation of Masticatory Performance by mixing ability of Hubba Bubba chewing gum.

The sample of 84 patients consisting of 42 cases and 42 controls. The patients will be re-evaluated at 2 and 3 months follow up for clinical periodontal parameters, masticatory performance and psychological distress.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with age group 30-50 years diagnosed with stage III/IV generalized periodontitis.
* Presence of minimum 20 teeth (Eichner group A1, A2, A3) excluding third molars.

Exclusion Criteria:

* Systemic diseases that may affect periodontal disease progression or outcome of treatment (diabetes, autoimmune diseases)
* Systemic diseases that may affect masticatory ability of the patient (sarcopenia, TMJ disorders, Xerostomia, Acute Pulpitis)
* Periodontal treatment within the 6 months
* Patients wearing orthodontic appliances
* Any diagnosed psychiatric disorder
* Antibiotic use within the previous 3 months
* Steroid, immunosuppressive and psychiatric drug use
* Pregnant and lactating women
* History of menopause
* Smoking or substance abuse

Ages: 30 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 92 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-09-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Masticatory performance | Baseline, 2 months, 3 months
  Objective Masticatory Performance will be evaluated using colour mixing ability of a chewing gum, through optoelectronic analysis using a software. Subjective masticatory performance will be calculated using The Quality of Masticatory Function questionnaire which consists of 29 questions related to frequency and difficulty of chewing different types of foods in the previous 2 weeks.
Hospital Anxiety and Depression Scale 14 | Baseline, 2 months, 3 months
  The HADS constitutes 14 items grouped into two subscales: "anxiety subscale" (HADS-A), as well as "depression subscale" (HADS-D). The responses to the items are graded from 0 (absence of manifestations) to 3 (severe manifestations). Scores are summated to yield the total score, and greater scores indicate more severe anxiety, as well as depressive indications. DASS-21 measures emotional distress in three subcategories of depression (e.g., loss of self-esteem/incentives and depressed mood), anxiety (e.g., fear and anticipation of negative events), and stress (e.g., persistent state of over arousal and low frustration tolerance). It is a self-reporting questionnaire with 21 items (seven items for each category) based on a four-point rating scale. Higher score represents more severe emotional distress.
Depression Anxiety and Stress Scale 21 | Baseline, 2 months, 3 months
  DASS-21 measures emotional distress in three subcategories of depression (e.g., loss of self-esteem/incentives and depressed mood), anxiety (e.g., fear and anticipation of negative events), and stress (e.g., persistent state of over arousal and low frustration tolerance). It is a self-reporting questionnaire with 21 items (seven items for each category) based on a four-point rating scale. Higher score represents more severe emotional distress.

SECONDARY OUTCOMES:
Pocket Probing Depth | Baseline, 2 months, 3 months
  The probe UNC 15 will be inserted with a firm, gentle pressure to the bottom of the pocket and maintained parallel to the vertical axis of the tooth. Measurements will be noted at 6 sites of involved tooth - mesio-buccal, mid-buccal, disto-buccal, mesio-lingual, mid-lingual, disto-lingual.
Clinical attachment level | Baseline, 2 months, 3 months
  Clinical Attachment Level will be measured as a distance between from the base of the clinical pocket and the cemento-enamel junction (CEJ). Measurements will be made at 6 sites of involved tooth.

CONTACTS AND LOCATIONS:
Overall Officials: Janvi Janvi, BDS, Principal Investigator — PGIDS Rohtak
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No